CLINICAL TRIAL: NCT04109456
Title: A Phase Ib, Open-label Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antitumor Activities of IN10018 as Monotherapy and Combination Therapy in Subjects With Metastatic Melanoma
Brief Title: IN10018 Monotherapy and Combination Therapy for Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InxMed (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IN10018-004-01
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Melanoma
Keywords: uveal; NRAS
MeSH Terms: conditions — Melanoma | interventions — cobimetinib; atezolizumab

STUDY DESIGN:
Intervention Model Description: The safety and tolerability of IN10018 monotherapy (Part 1) will be assessed firstly. Other dose levels may be explored if necessary.
  and then the safety and tolerability of IN10018 in combination with Cobimetinib (Part 2) will be evaluated.
  the safety and tolerability of IN10018 in combination with Cobimetinib and Atezolizumab (Part 3) will be evaluated .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1, Monotherapy Arm (Experimental): The safety and tolerability of IN10018 monotherapy will be assessed. Other dose levels may be explored if necessary.
  Interventions: Drug: IN10018
- Part 2, Combination Arm (Experimental): The safety and tolerability of IN10018 in combination with Cobimetinib will be assessed. Other dose levels may be explored if necessary.
  A modified 3+3 design will be used.
  Interventions: Drug: IN10018; Drug: Cobimetinib
- Part 3, Combination Arm (Experimental): The safety and tolerability of IN10018 in combination with Cobimetinib and Atezolizumab will be assessed.
  Interventions: Drug: IN10018; Drug: Cobimetinib; Biological: Atezolizumab

INTERVENTIONS:
Drug: IN10018 — 100 mg or 50mg, orally once daily continuously;
  Other Names: BI 853520
Drug: Cobimetinib — 60mg , orally once daily from day 1 to day 21 in a 28-day cycle
  Other Names: Cotellic
  Arms: Part 2, Combination Arm; Part 3, Combination Arm
Biological: Atezolizumab — biweekly 840 mg dose will be used in this study starting from Cycle 2.
  Arms: Part 3, Combination Arm

SUMMARY:
This is a phase Ib, open label clinical study to evaluate the safety, tolerability, PK and antitumor activities of IN10018 as monotherapy and in combination with cobimetinib in subjects with metastatic uveal melanoma and NRAS-mutant metastatic melanoma.

DETAILED DESCRIPTION:
Subjects with metastatic uveal melanoma (UM) or with NRAS-mutant metastatic melanoma will be enrolled.

IN10018 will be assessed firstly as monotherapy（Part 1）, then in combination with cobimetinib (Part 2) and in combination with cobimetinib and Atezolizumab (Part 3).

ELIGIBILITY:
Key Inclusion Criteria:

1. Ability to understand and willingness to sign informed consent(s).
2. Male or female subjects ≥ 18 years at the time of signing informed consent.
3. Histologically or cytologically confirmed metastatic melanoma with subtypes limited to:

   1. Metastatic uveal melanoma, or
   2. Metastatic NRAS-mutant melanoma harboring an NRAS activating mutations of Q61, G12, or G13 mutation per local laboratory (including local reference laboratory) results.
4. Requirements for previous therapy:

   1. Uveal melanoma: Either be treatment naïve or have failed the most recent therapy for metastatic disease, or
   2. NRAS-mutant melanoma: Either be ineligible for standard of care due to the presence of various comorbidities or have failed the most recent therapy such as immunotherapy for metastatic disease.
   3. Have failed immunotherapy therapy (anti-PD-1 or anti-PD-L1) alone or in combination with other agents for metastatic disease either with no initial response or disease progression after an initial response. (Part 3)
   4. Received a minimum of two cycles of anti-PD-1/PD-L1 therapy. (Part 3)
5. Consent to undergo tumor biopsies of accessible lesions, before and during treatment and at radiographic progression, for biomarker analyses (site dependent).
6. At least one measurable lesion can be accurately measured per RECIST 1.1 by investigator.
7. ECOG performance status of 0 or 1.
8. Life expectancy of at least 3 months as assessed by investigator.
9. Availability of fresh tumor tissue and/or archival tumor tissue at Screening if agreed by subjects.
10. Must have recovered from all AEs due to previous therapies to ≤ Grade 1 (CTCAE 5.0) or stable status as assessed by investigator.
11. Adequate bone marrow, liver, renal, and coagulation function within 5 days prior to first dose of study treatment.
12. A male subject must agree to use contraception as detailed in Appendix 4 of this protocol during the treatment period and through 30 days after the last dose of study treatment and must refrain from donating sperm during this period.
13. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 4. OR
    2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 4 during the treatment period and through 30 days after the last dose of study treatment.

Key Exclusion Criteria:

1. Has had major surgery or significant traumatic injury within 28 days prior to first dose of study treatment, or anticipation of the need for major surgery during study treatment.
2. Has received prior systemic, intrahepatic, or sphere anticancer therapy including investigational agents within 14 days or less than 5 half-lives (whichever is shorter) of chemotherapy or targeted therapy, or within 28 days of immunotherapy, prior to first dose of study treatment.
3. Has received prior radiotherapy or radioactive chemotherapy within 14 days prior to first dose of study treatment.
4. Has received prior treatment of any FAK inhibitor (Parts 1, 2 and 3), or prior treatment of any MEK inhibitor (Parts 2 and 3 only).
5. Has a known previous or concurrent cancer that is distinct in primary site or histology from current melanoma within 3 years prior to first dose of study treatment, except for curatively treated cancers such as cervical carcinoma in situ and indolent cancers with very low likelihood of relapse or progress per investigator judgement.
6. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
7. Diabetes mellitus, insulin dependent and non-insulin dependent with HBA1C > 6.5%, microalbuminuria > 150 mg (24-h collection), and CrCL of < 45ml/min with an adequate 24-hour urine collection.
8. Prior history of Alport syndrome.
9. Recent medical history (with the last 1-year) of acute renal injury, Goodpasture's Syndrome, IgA nephropathy, focal segmental glomerulosclerosis, nephrotic syndrome, parenteral drug abuse, recurrent pyelonephritis, systemic lupus erythematosus, uncontrolled hypertension, vasculitis, and chronic illnesses with potential underlying glomerular renal disease.
10. Has contraindications to anti-PD-1 or anti-PD-L1 immunotherapy (Part 3).
11. Has received prior treatment with anti-PD-1, anti-PD-L1, or anti-CTLA4 immunotherapy and was discontinued for significant immunotherapy-related adverse events (Part 3).
12. Current treatment with anti-viral therapy for HBV (Part 3).
13. Prior allogeneic stem cell or solid organ transplantation.
14. Active tuberculosis
15. Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina (Part 3).
16. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions: Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study. (Part 3).
17. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on previous chest computed tomography (CT) scan.
18. Has a history of major cardiovascular, cerebrovascular, or thromboembolic diseases (e.g., congestive heart failure, acute myocardial infarction, unstable angina, atrial fibrillation, ventricular tachyarrhythmia, uncontrolled hypertension, stroke, transient ischemic attack, deep vein thrombosis or pulmonary embolism) within 6 months before first dose of study treatment, or has any of the following abnormality:

    * QTc interval > 480 msec (Fridericia formula), (patients with right bundle branch block is not required to have QTc if the block is stable and assessed as not clinically significant by the PI),
    * Left ventricular ejection fraction (LVEF) < 50%,
    * Arrhythmia with clinical significance, or
    * Other heart diseases with clinical significance.
19. History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment/ central serous chorioretinopathy (CSCR), retinal vein occlusion (RVO), neovascular macular degeneration, or uncontrolled glaucoma with intra-ocular pressures >21 mmHg in the eye(s) unaffected by melanoma. (Parts 2 and 3)
20. Has known uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage prior to the first dose of study treatment.
21. Has malabsorption syndrome or inability to take oral drugs.
22. Has clinically significant gastrointestinal abnormalities including uncontrolled gastrointestinal inflammatory lesions (Crohn's disease, or ulcerative colitis in active or uncontrolled gastrointestinal bleeding).
23. Known allergy or hypersensitivity to IN10018 cobimetinib and/or atezolizumab, or their ingredients.
24. Has had an active infection requiring systemic therapy within 14 days prior to the first dose of study treatment.
25. Has known human immunodeficiency virus (HIV) infection.
26. Has known active Hepatitis B or Hepatitis C virus infection.
27. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
28. Has a known psychiatric or substance abuse disorder that would interfere with the subject's ability to cooperate with the requirements of the study.
29. Has had used below CYP3A inhibitors/inducers and P-gp inhibitors within 14 days prior to first dose of study treatment, or anticipation of the need to use them during study treatment:

    * Part 1: Strong CYP3A inhibitors/inducers and P-gp inhibitors are prohibited at least 14 days prior to initiation of and during study treatment.
    * Parts 2 and 3: Moderate and Strong CYP3A inhibitors/inducers and P-gp inhibitors are prohibited at least 14 days prior to initiation of and during study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of IN10018 monotherapy | The first 21-day cycle
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment
Safety and tolerability of IN10018 in combination with cobimetinib | The first 28-day cycle
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment
Safety and tolerability of IN10018 in combination with cobimetinib and atezolizumab | All treatment period
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment

SECONDARY OUTCOMES:
Pharmacokinetics (PK) : Cmax | Cycle 1 and Cycle 3
  Peak Plasma Concentration (Cmax)
Pharmacokinetics (PK) : AUC | Cycle 1 and Cycle 3
  Area under the plasma concentration versus time curve (AUC)
Pharmacokinetics (PK) : tmax | Cycle 1 and Cycle 3
  Time to Cmax (tmax)
Pharmacokinetics (PK) : t1/2 | Cycle 1 and Cycle 3
  Elimination half-life (t1/2)
Pharmacokinetics (PK) : CL/F | Cycle 1 and Cycle 3
  apparent clearance (CL/F)
Pharmacokinetics (PK) : Vd | Cycle 1 and Cycle 3
  Apparent volume of distribution(Vd)
Overall Response Rates using RECiST1.1 criteria | 1 year
  Proportion of participants with (complete response, partial response, stable disease, progressive disease) in all 3 parts
Disease Control Rate using RECiST1.1 criteria | 1 year
  Proportion of subjects who have disease control (CR, PR or stable disease (SD)) in all 3 parts
duration of response (DOR) | 1 year
  For subjects who demonstrate CR or PR, DOR is defined as the time from first evidence of CR or PR until PD or death due to any cause, whichever occurs first in all 3 parts
progression free survival (PFS) | 1 year
  PFS is defined as the time from the first day of study treatment to the first disease progression or death due to any cause, whichever occurs first in all 3 parts
overall survival (OS) | 1 year
  OS is defined as the time from the first day of study treatment to death due to any cause in all 3 parts

OTHER OUTCOMES:
To explore potential predictive biomarkers | through study completion, an average of 5 year
  in all 3 parts

CONTACTS AND LOCATIONS:
Overall Officials: Eddie Xing, Dr., Study Director — InxMed Shanghai
Locations (8):
- United States (5):
  - Sylvester Comprehensive Cancer Center., Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - MD Anderson, Houston, Texas
- Australia (3):
  - St Vincent Hospital Sydney, Sydney, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No